CLINICAL TRIAL: NCT02023125
Title: An Open-Label, Two-Group Study to Investigate the Effect of Food (Group 1) and Esomeprazole (Group 2) on the Single Oral Dose Pharmacokinetics of RO5424802 in Healthy Subjects
Brief Title: A Study Investigating the Effect of Food and Esomeprazole on the Single Oral Dose Pharmacokinetics of Alectinib (RO5424802) in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP28991
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — alectinib; Esomeprazole

ARMS (3):
- Group 1: Treatment A first, then Treatment B (Experimental): Treatment A (Fasted Treatment): Following an overnight fast of at least 10 hours, a single 600-mg oral dose of alectinib will be administered. Treatment B (Fed Treatment): Following an overnight fast of at least 10 hours, participants will start a high-fat, high-calorie meal 30 minutes prior to study drug administration; study participants should eat this meal in 30 minutes or less. The single 600-mg oral dose of alectinib will be administered 30 minutes after the start of the meal. Each period will be separated by at least 10 days.
  Interventions: Drug: Alectinib; Other: High Fat and Calorie Meal
- Group 1: Treatment B first, then Treatment A (Experimental): Treatment B (Fed Treatment): Following an overnight fast of at least 10 hours, participants will start a high-fat, high-calorie meal 30 minutes prior to study drug administration; study participants should eat this meal in 30 minutes or less. The single 600-mg oral dose of alectinib will be administered 30 minutes after the start of the meal. Treatment A (Fasted Treatment): Following an overnight fast of at least 10 hours, a single 600-mg oral dose of alectinib will be administered. Each period will be separated by at least 10 days.
  Interventions: Drug: Alectinib; Other: High Fat and Calorie Meal
- Group 2: Alectinib Alone, Alectinib + Esomeprazole (Experimental): Period 1 (Days 1 to 10): Following an overnight fast of at least 10 hours, participants will start a standardized meal and should consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib will be administered 30 minutes after the start of the meal on Day 1 of Period 1. Period 2 (Days 11 to 20): Participants will receive oral esomeprazole 40 mg once daily for 6 days (Days 11-16) in the morning after an overnight fast of at least 10 hours, and at least 1 hour before a regular breakfast; On Day 16, following an overnight fast of at least 10 hours, a single oral dose of 40 mg esomeprazole will be administered 1.5 hours prior to the start of a standardized meal. Following a standardized meal, a single oral 600 mg dose of alectinib will then be administered.
  Interventions: Drug: Alectinib; Drug: Esomeprazole; Other: Standard Meal

INTERVENTIONS:
Drug: Alectinib — A single 600-mg oral dose of alectinib will be administered in a fasted or fed condition.
  Other Names: RO5424802
Drug: Esomeprazole — Esomeprazole 40 mg will be administered orally once daily for 6 days prior to alectinib administration.
  Arms: Group 2: Alectinib Alone, Alectinib + Esomeprazole
Other: High Fat and Calorie Meal — High fat and calorie meal served prior to alectinib administration
  Arms: Group 1: Treatment A first, then Treatment B; Group 1: Treatment B first, then Treatment A
Other: Standard Meal — Standard meal served prior to alectinib administration
  Arms: Group 2: Alectinib Alone, Alectinib + Esomeprazole

SUMMARY:
This two-group study will investigate the effect of food (Group 1) and esomeprazole (Group 2) on the single oral dose pharmacokinetics of alectinib in healthy volunteers.

Participants in Group 1 will be randomly assigned to a two period treatment sequence (AB or BA) in which they will receive a single, oral dose of alectinib per period separated by at least 10 days. Each participant will receive single, oral doses alectinib given under fasted conditions (Treatment A) or following the ingestion of a high fat, high calorie meal (Treatment B) as determined by their assigned sequence.

Participants in Group 2 will be given a single, oral dose of alectinib following a standard meal. After a washout period of at least 10 days, they will receive an oral dose of esomeprazole (40 mg) once daily for 6 days. On the 6th day of esomeprazole administration, a single, oral dose alectinib will be given after ingestion of a standard meal.

In all groups, pharmacokinetics will be assessed in the 4 days following alectinib administration.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 to 32 kilogram per square meter (kg/m^2)
* Healthy male and female participants. Healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead electrocardiogram (ECG), hematology, blood chemistry, serology and urinalysis
* Female participants must be surgically sterile or post-menopausal for the past year confirmed by a blood follicle stimulating hormone (FSH) test for females without hormone replacement therapy (HRT)
* Male participants must be willing to use effective contraception, as defined by the protocol, throughout the study and for 3 months after last drug administration
* Willing to abstain from xanthine-containing beverages or food (coffee, tea, cola, chocolate, and "energy drinks") use from 72 hours prior to admission to the study clinic until discharge
* Willing to abstain from consuming grapefruit, pomelo, star fruit, or Seville orange containing products from 7 days prior to first dose of study medication through discharge
* Willing to avoid prolonged sun exposure while taking alectinib and through follow-up. Participants should also be advised to use a broad spectrum sun screen and lip balm of at least sun protection factor (SPF) > 30 to help protect against potential sunburn
* Group 2 participants should be H. Pylori negative via breath test

Exclusion Criteria:

* Pregnant or breastfeeding women, males with female partners who are pregnant or breastfeeding, or women of childbearing potential.
* Positive test for drugs of abuse, alcohol or cotinine test at screening or prior to admission to the study unit
* Suspicion of regular consumption of drug(s) of abuse including marijuana.
* Current smokers or participants who have discontinued smoking less than six months prior to first dosing. Participants should avoid smoky environments for at least 1 weeks prior to each cotinine test
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 10 grams of alcohol). Alcohol consumption will be prohibited 72 hours prior to admission to the study clinic and throughout the entire study until discharge
* Participants with any risk factors or family history for QT/QTcF prolongation or ECG abnormalities or any abnormality in the ECG that, in the opinion of the investigator, increases the risk of participating in the study
* Confirmed systolic blood pressure (SBP) greater than 140 millimeter of mercury (mmHg) or less than 90 mmHg or diastolic blood pressure (DBP) greater than 90 mmHg or less than 45 mmHg at screening, admission to the study center or prior to dosing.
* Notable resting bradycardia (mean pulse rate < 45 beats per minute [bpm]) or tachycardia (mean pulse rate > 90 bpm)
* Use of any medications (prescription or over-the-counter) within 2 weeks or 5 half-lives (whichever is longer) before the first dose of the study medication with the exception of acetaminophen up to 2 g per day up to 48 hours prior to dosing, not to exceed 4 g total during the week prior to dosing
* Use of any herbal supplements or any metabolic inducers within 4 weeks or 5 half-lives (whichever is longer) before the first dose of study medication, including but not limited to the following drugs: rifampin, rifabutin, glucocorticoids, carbamazepine, phenytoin and phenobarbital
* Strenuous activity, sunbathing or contact sports are not allowed from 4 days prior to entry into the clinical site and for the duration of the study until follow-up
* Participation in an investigational drug or device study within 45 days or 5 half-lives (whichever is longer) or 6 months for biologic therapies prior to first dosing
* Donation of blood over 450 mL within 45 days prior to screening
* Regular use of antacids, Histamine 2 (H2) receptor blockers, proton pump inhibitors (PPIs) or any medications which may alter the normal gastric environment and/or motility. No use of such medications within 2 weeks prior to first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Treatment A First, Then Treatment B: Treatment A (Fasted Treatment): Following an overnight fast of at least 10 hours, a single 600 milligrams (mg) oral dose of alectinib was administered. Treatment B (Fed Treatment): Following an overnight fast of at least 10 hours, participants started a high-fat, high-calorie meal 30 minutes prior to study drug administration and were to consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal. Each period was separated by at least 10 days.
- Group 1: Treatment B First, Then Treatment A: Treatment B (Fed Treatment): Following an overnight fast of at least 10 hours, participants started a high-fat, high-calorie meal 30 minutes prior to study drug administration and were to consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal. Treatment A (Fasted Treatment): Following an overnight fast of at least 10 hours, a single 600-mg oral dose of alectinib was administered. Each period was separated by at least 10 days.
- Group 2: Alectinib Alone, Alectinib + Esomeprazole: Period 1 (Days 1 to 10): Following an overnight fast of at least 10 hours, participants started a standardized meal and were to consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal on Day 1 of Period 1. Period 2 (Days 11 to 20): Participants received oral esomeprazole 40 mg once daily for 6 days (Days 11-16) in the morning after an overnight fast of at least 10 hours, and at least 1 hour before a regular breakfast; On Day 16, following an overnight fast of at least 10 hours, a single oral dose of 40 mg esomeprazole was administered 1.5 hours prior to the start of a standardized meal. Following a standardized meal, a single oral 600 mg dose of alectinib was then administered.
Period: Period 1
Arm/Group | Group 1: Treatment A First, Then Treatment B | Group 1: Treatment B First, Then Treatment A | Group 2: Alectinib Alone, Alectinib + Esomeprazole
Started | 9 | 9 | 24
Completed | 9 | 9 | 24
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Group 1: Treatment A First, Then Treatment B | Group 1: Treatment B First, Then Treatment A | Group 2: Alectinib Alone, Alectinib + Esomeprazole
Started | 9 | 9 | 24
Completed | 9 | 9 | 24
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Group 1: Treatment A First, Then Treatment B | Group 1: Treatment B First, Then Treatment A | Group 2: Alectinib Alone, Alectinib + Esomeprazole
Started | 9 | 9 | 24
Completed | 9 | 9 | 24
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all participants who received at least 1 dose of study drug and had at least 1 after dosing safety assessment.
Groups:
- Group 1 (Treatment Sequence AB or BA): Participants in Group 1 were randomly assigned to a two period treatment sequence (AB or BA) in which they received a single, oral dose of 600 mg of alectinib per period separated by at least 10 days. Each participant received single, oral doses alectinib given under fasted conditions (Treatment A) or following the ingestion of a high fat, high calorie meal (Treatment B) as determined by their assigned sequence.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Treatment Sequence AB or BA) | Group 2: Alectinib Alone, Alectinib + Esomeprazole | Total
Number analyzed (Participants) | 18 | 24 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (8.50) | 35.4 (8.30) | 35.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Alectinib: Group 1
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: Pharmacokinetic (PK) Analysis Population [Group 1] consisted of all participants who received both scheduled doses of Alectinib, and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Group 1: Treatment A (Fasted Treatment): Following an overnight fast of at least 10 hours, a single 600-mg oral dose of alectinib was administered.
- Group 1: Treatment B (Fed Treatment): Following an overnight fast of at least 10 hours, participants started a high-fat, high-calorie meal 30 minutes prior to study drug administration and were to consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal.
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
nanograms per milliliter (ng/mL) | 103 (41.1) | 270 (86.4)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); Analysis of variance (ANOVA) was applied to the log-transformed PK parameter and then back transformed to provide geometric least square mean ratios (Treatment B/Treatment A) and confidence intervals (CIs); Test type: Superiority or Other; Geometric Least Square Mean Ratio = 270, 90% CI 2-sided [228 to 320] — The reported values are percentages of geometric least square mean ratio

2. Primary Outcome: Cmax of Alectinib: Group 2
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours post alectinib dose in each treatment period
Population: PK Analysis Population [Group 2] consisted of all participants who received both scheduled doses of Alectinib, and provided adequate PK assessments.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 2: Period 1 (Alectinib Alone): Period 1 (Days 1 to 10): Following an overnight fast of at least 10 hours, participants started a standardized meal and were to consume the meal in 30 minutes or less. The single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal on Day 1 of Period 1.
- Group 2: Period 2 (Alectinib + Esomeprazole): Period 2 (Days 11 to 20): Participants received oral esomeprazole 40 mg once daily for 6 days (Days 11-16) in the morning after an overnight fast of at least 10 hours, and at least 1 hour before a regular breakfast; On Day 16, following an overnight fast of at least 10 hours, a single oral dose of 40 mg esomeprazole was administered 1.5 hours prior to the start of a standardized meal. Following a standardized meal, a single oral 600 mg dose of alectinib was then administered.
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
ng/mL | 169 (47.3) | 196 (54.7)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); ANOVA was applied to the log-transformed PK parameter and then back transformed to provide geometric least square mean ratios (Alectinib + Esomeprazole/Alectinib Alone) and CIs; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 116, 90% CI 2-sided [103 to 132] — The reported values are percentages of geometric least square mean ratio

3. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of Alectinib: Group 1
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
hours*nanograms per milliliter (h*ng/mL) | 1900 (665) | 5480 (1800)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); ANOVA was applied to the log-transformed PK parameter and then back transformed to provide geometric least square mean ratios (Treatment B/Treatment A) and CIs; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 292, 90% CI 2-sided [258 to 329] — The reported values are percentages of geometric least square mean ratio

4. Primary Outcome: AUC0-inf of Alectinib: Group 2
Description: as for outcome 3
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
h*ng/mL | 3180 (876) | 3940 (1310)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 122, 90% CI 2-sided [109 to 136] — The reported values are percentages of geometric least square mean ratio

5. Secondary Outcome: Cmax of RO5468924: Group 1
Description: RO5468924 is M4 metabolite of alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
ng/mL | 37.5 (20.7) | 126 (31.9)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 377, 90% CI 2-sided [303 to 468] — The reported values are percentages of geometric least square mean ratio

6. Secondary Outcome: Cmax of RO5468924: Group 2
Description: RO5468924 is M4 metabolite of alectinib.
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
ng/mL | 72.1 (28.8) | 72.1 (26.4)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 102, 90% CI 2-sided [87.0 to 119] — The reported values are percentages of geometric least square mean ratio

7. Secondary Outcome: AUC0-inf of RO5468924: Group 1
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf). RO5468924 is M4 metabolite of alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
h*ng/mL | 1140 (497) | 3480 (758)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 328, 90% CI 2-sided [276 to 389] — The reported values are percentages of geometric least square mean ratio

8. Secondary Outcome: AUC0-inf of RO5468924: Group 2
Description: as for outcome 7
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
h*ng/mL | 1860 (639) | 2050 (713)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 110, 90% CI 2-sided [96.3 to 126] — The reported values are percentages of geometric least square mean ratio

9. Secondary Outcome: Metabolite/Parent Ratio for AUC0-inf: Group 1
Description: AUC (0-inf) = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0 - t) plus AUC (t - inf). RO5468924 is M4 metabolite of alectinib. The ratio is molecular weight adjusted.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
ratio | 0.610 (0.07) | 0.686 (0.08)

10. Secondary Outcome: Metabolite/Parent Ratio for AUC0-inf: Group 2
Description: as for outcome 9
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
ratio | 0.548 (0.05) | 0.607 (0.08)

11. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Alectinib: Group 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
h*ng/mL | 1780 (648) | 5360 (1750)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 306, 90% CI 2-sided [269 to 348] — The reported values are percentages of geometric least square mean ratio

12. Secondary Outcome: AUClast of Alectinib: Group 2
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
h*ng/mL | 3050 (867) | 3790 (1280)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 122, 90% CI 2-sided [110 to 136] — The reported values are percentages of geometric least square mean ratio

13. Secondary Outcome: AUClast of RO5468924: Group 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). RO5468924 is M4 metabolite of alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
h*ng/mL | 1030 (491) | 3290 (715)
Statistical Analysis 1: Comparison: Group 1: Treatment A (Fasted Treatment) vs Group 1: Treatment B (Fed Treatment); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 349, 90% CI 2-sided [288 to 422] — The reported values are percentages of geometric least square mean ratio

14. Secondary Outcome: AUClast of RO5468924: Group 2
Description: as for outcome 13
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
h*ng/mL | 1750 (617) | 1920 (685)
Statistical Analysis 1: Comparison: Group 2: Period 1 (Alectinib Alone) vs Group 2: Period 2 (Alectinib + Esomeprazole); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Geometric Least Square Mean Ratio = 109, 90% CI 2-sided [95.3 to 126] — The reported values are percentages of geometric least square mean ratio

15. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Alectinib: Group 1
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
hours | 4.00 [2.00 to 8.00] | 8.00 [6.00 to 12.0]

16. Secondary Outcome: Tmax of Alectinib: Group 2
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Median (Full Range); unit: hours
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
hours | 6.00 [4.00 to 10.0] | 6.00 [4.00 to 10.0]

17. Secondary Outcome: Tmax of RO5468924: Group 1
Description: RO5468924 is M4 metabolite of alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
hours | 8.00 [4.02 to 12.0] | 10.0 [6.00 to 12.0]

18. Secondary Outcome: Tmax of RO5468924: Group 2
Description: RO5468924 is M4 metabolite of alectinib.
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Median (Full Range); unit: hours
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
hours | 6.02 [6.00 to 12.0] | 8.00 [6.00 to 12.0]

19. Secondary Outcome: Terminal Half-life (t1/2) of Alectinib: Group 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
hours | 23.4 (13.7) | 17.7 (5.12)

20. Secondary Outcome: t1/2 of Alectinib: Group 2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
hours | 20.4 (9.33) | 20.4 (7.56)

21. Secondary Outcome: t1/2 of RO5468924: Group 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. RO5468924 is M4 metabolite of alectinib.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment period
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
hours | 29.4 (7.05) | 22.7 (3.27)

22. Secondary Outcome: t1/2 of RO5468924: Group 2
Description: as for outcome 21
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Group 2: Period 2 (Alectinib + Esomeprazole): Period 2 (Day 16): Participants started the standardized meal 30 minutes prior to administration of alectinib. Participants were to consume this meal in 30 minutes or less. A single 600-mg oral dose of alectinib was administered 30 minutes after the start of the meal. Period 2 (Days 11 to 20): From Days 11 to 15 esomeprazole 40 mg was administered orally once daily in the morning after an overnight fast of at least 10 hours, and at least 1 hour before a regular breakfast; On Day 16, following an overnight fast of at least 10 hours, a single oral dose of 40-mg esomeprazole was administered 1.5 hours prior to the start of a standardized meal.
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
hours | 25.0 (4.56) | 25.4 (5.06)

23. Secondary Outcome: Apparent Oral Clearance (CL/F) for Alectinib: Group 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: Liters per hour (L/h)
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
Liters per hour (L/h) | 357 (136) | 120 (38.1)

24. Secondary Outcome: CL/F for Alectinib: Group 2
Description: as for outcome 23
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
L/h | 206 (72.5) | 170 (61.0)

25. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Alectinib: Group 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed.
Time Frame: Predose (0 hours) and at 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours after dosing in each treatment arm
Population: PK Analysis Population [Group 1]
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment)
Number analyzed (Participants) | 18 | 18
Liters | 11800 (7200) | 3060 (1290)

26. Secondary Outcome: Vz/F for Alectinib: Group 2
Description: as for outcome 25
Time Frame: as for outcome 2
Population: PK Analysis Population [Group 2]
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Number analyzed (Participants) | 24 | 24
Liters | 5930 (2950) | 4890 (2070)

ADVERSE EVENTS:
Time Frame: Day 1 up to 7 to 10 days after last dose of alectinib (Cohort 1: maximum up to 18 to 21 days; Cohort 2: maximum up to 23 to 26 days)
Description: Safety Analysis Set.
Groups:
- Group 2: Period 2 (Esomeprazole Alone): Period 2: From Days 11 to 15 esomeprazole 40 mg was administered orally once daily in the morning after an overnight fast of at least 10 hours, and at least 1 hour before a regular breakfast.
Arm/Group | Group 1: Treatment A (Fasted Treatment) | Group 1: Treatment B (Fed Treatment) | Group 2: Period 1 (Alectinib Alone) | Group 2: Period 2 (Esomeprazole Alone) | Group 2: Period 2 (Alectinib + Esomeprazole)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 8/18 | 8/18 | 5/24 | 3/24 | 4/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Treatment A (Fasted Treatment) (N=18) | Group 1: Treatment B (Fed Treatment) (N=18) | Group 2: Period 1 (Alectinib Alone) (N=24) | Group 2: Period 2 (Esomeprazole Alone) (N=24) | Group 2: Period 2 (Alectinib + Esomeprazole) (N=24)
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1
Lip dry (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0
Influenza-like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Application site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.